CLINICAL TRIAL: NCT04788264
Title: A Pilot Study to Assess Feasibility of a Clinically Significant Increase in Physical Activity in Patients With Head and Neck Cancer Undergoing Active Treatment
Brief Title: Exercise Training and Behavioral Modification for the Improvement of Physical Activity in Head and Neck Cancer Patients Undergoing Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20D.775; JT 15554 (Other: JeffTrial Number); 108 27000 908059 (Other Grant/Funding Number: Population Science Cancer Research Fund)
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Carcinoma; Hypopharyngeal Carcinoma; Laryngeal Carcinoma; Maxillary Sinus Carcinoma; Oral Cavity Carcinoma; Oropharyngeal Carcinoma; Paranasal Sinus Carcinoma; Sinonasal Carcinoma; Stage I Laryngeal Cancer AJCC v8; Stage II Laryngeal Cancer AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVC Laryngeal Cancer AJCC v8; Lung Carcinoma
MeSH Terms: conditions — Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Maxillary Sinus Neoplasms; Mouth Neoplasms; Oropharyngeal Neoplasms; Paranasal Sinus Neoplasms; Lung Neoplasms | interventions — Referral and Consultation; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (exercise training, behavior modification) (Experimental): Beginning 1 week prior to start of intervention, patients receive a Fitbit to monitor physical activity for 13 weeks. Patients receive consultation and personalized exercise prescription from a physical therapist at baseline, and attend exercise training sessions with a physical therapist during weeks 1, 3, 6, 9, and 12. Patients also attend behavior modification sessions with a behavioral therapist that focus on goal setting and healthy behavior changes during weeks 2, 4, 5, 7, 8, 10, and 11.
  Interventions: Other: Medical Device Usage and Evaluation; Other: Consultation; Other: Exercise Intervention; Behavioral: Behavioral Intervention; Other: Questionnaire Administration; Other: Quality of Life Assessment
- Arm II (Fitbit, consultation) (Active Comparator): Patients receive a Fitbit to monitor physical activity for 12 weeks. Patients also receive consultation from a physical therapist to assess physical performance at weeks 1, 6, and 12.
  Interventions: Other: Medical Device Usage and Evaluation; Other: Consultation; Other: Questionnaire Administration; Other: Quality of Life Assessment

INTERVENTIONS:
Other: Medical Device Usage and Evaluation — Receive Fitbit
Other: Consultation — Receive consultation from a physical therapist
  Other Names: Consult
Other: Exercise Intervention — Attend exercise training sessions
  Arms: Arm I (exercise training, behavior modification)
Behavioral: Behavioral Intervention — Attend sessions with a behavioral therapist
  Other Names: Behavior Conditioning Therapy
  Arms: Arm I (exercise training, behavior modification)
Other: Questionnaire Administration — Ancillary studies
Other: Quality of Life Assessment — Ancillary studies

SUMMARY:
This clinical trial evaluates the tolerability of a physical activity program in head and neck cancer patients who are undergoing cancer treatment. The goal of this trial is to give patients exercises prescribed by a physical therapist that they are able to complete regularly at home. Increasing physical activity may help patients reduce fatigue, improve mood, increase physical performance, and decrease joint pain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the changes in physical activity between the control and intervention groups of patients with head and neck or lung cancer at 6-weeks and 12-weeks, compared to baseline.

SECONDARY OBJECTIVES:

I. To demonstrate the feasibility, engagement, retention, and acceptability of physical activity promotion (intervention) in patients with head and neck or lung cancer.

II. To calculate the effect sizes for the differences between the control and intervention in daily changes in psychosocial outcomes at 6-weeks and 12-weeks, compared to baseline.

EXPLORATORY OBJECTIVE:

I. To calculate the effect sizes for the differences between the control and intervention in changes in immunomodulatory, metabolic and aging biomarkers at 6-weeks and 12-weeks, compared to baseline.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Beginning 1 week prior to start of intervention, patients receive a Fitbit to monitor physical activity for 13 weeks. Patients receive consultation and personalized exercise prescription from a physical therapist at baseline, and attend exercise training sessions with a physical therapist during weeks 1, 3, 6, 9, and 12. Patients also attend behavior modification sessions with a behavioral therapist that focus on goal setting and healthy behavior changes during weeks 2, 4, 5, 7, 8, 10, and 11.

ARM II: Patients receive a Fitbit to monitor physical activity for 12 weeks. Patients also receive consultation from a physical therapist to assess physical performance at weeks 1, 6, and 12.

After completion of study intervention, patients are followed up at 30 days.

EXPLORATORY OBJECTIVE:

I. To demonstrate the difference in the magnitude of physical activity improvements between the immunotherapy and chemo-immunotherapy patients.

OUTLINE:

Beginning 1 week prior to start of intervention, patients receive a Fitbit to monitor physical activity for 13 weeks. Patients receive consultation and personalized exercise prescription from a physical therapist at baseline, and attend exercise training sessions with a physical therapist during weeks 1, 3, 6, 9, and 12. Patients also attend behavior modification sessions with a behavioral therapist that focus on goal setting and healthy behavior changes during weeks 2, 4, 5, 7, 8, 10, and 11.

After completion of study intervention, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with head and neck cancer including cancers of the sinuses, oral cavity, oropharynx, hypopharynx, or larynx (all stages); therapeutically eligible to receive at least three months of immunotherapy
* Medically cleared by oncologist to engage in aerobic and resistance exercise intervention
* 18 years of age or older
* Access to a smartphone and have an active wi-fi connection at home
* Able to read and/or to speak English
* Able to comprehend and sign a written informed consent (no cognitive decline)
* Women of reproductive potential must have a negative serum or urine pregnancy test within the week prior to starting therapy

Exclusion Criteria:

* Severe or unstable cardiopulmonary, metabolic, or renal disease as determined by the referring oncologist
* Unable to walk safely without physical assistance of another person
* Any condition that may limit the ability to comply with behavioral recommendations of the program
* Pregnant or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-28 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Change in Fitbit-recorded average steps (moderate and/or intensive) per day, each day | Baseline to 12 weeks after physical activity promotion
  Changes in physical activity of the intervention group at 6-weeks and 12-weeks, compared to baseline, using two-sample t-tests, respectively. Longitudinal models such as (non)linear mixed models or generalized estimating equation (GEE) models
Change in Fitbit-recorded average steps (moderate and/or intensive) per day, each day | Baseline to 12 weeks after physical activity promotion
  Changes in physical activity of the control group at 6-weeks and 12-weeks, compared to baseline, using two-sample t-tests, respectively. Longitudinal models such as (non)linear mixed models or generalized estimating equation (GEE) models
Change in Fitbit-recorded average active minutes (moderate and/or intensive) per day, each day | Baseline to 12 weeks after physical activity promotion
  time trend will be compared between control and intervention groups at 6-weeks and 12-weeks, compared to baseline, using two-sample t-tests, respectively. Longitudinal models such as (non)linear mixed models or generalized estimating equation (GEE) models

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No